CLINICAL TRIAL: NCT00847002
Title: A Pilot Randomized Trial of Flexitouch as an Adjunctive Treatment for Venous Ulcers
Brief Title: Flexitouch Treatment for Venous Ulcers
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of Enrollment
Sponsor: Tactile Systems Technology, Inc. (Industry)
Responsible Party: Sponsor
Organization: Tactile Medical (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FWFT07312007
Record Dates: First submitted 2009-02-18; First posted 2009-02-19 (Estimated); Results first posted 2012-07-25 (Estimated); Last update posted 2020-02-12 (Actual); Status verified 2020-01

CONDITIONS: Venous Ulcer
Keywords: Flexitouch system; FarrowWrap; venous stasis ulcer
MeSH Terms: conditions — Varicose Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Standard Wound Care (Active Comparator): Gentle wound ulcer cleansing with saline solution at each visit, maintaining moisture balance in the wound and periwound with appropriate dressings (e.g Acticoat, Aquacel Ag, or Mepilex Ag foam dressings), reminding subjects of importance of proper nutrition, leg elevation at rest and activity, including frequent ambulation and ankle range of motion exercises through the day. The FarrowWrap Classic device is applied over the dressing to achieve suitable compression pressures as an important component of the standard treatment.
  Interventions: Device: Standard Wound Care
- Flexitouch system with Standard Wound Care (Active Comparator): In addition to standard wound care, patients who have been randomized to this group will be provided a home Flexitouch unit. They will be given instructions to use it on a twice daily basis (FarrowWrap will be removed during the time they are using Flexitouch). The Flexitouch System works by applying dynamic low-pressure compression to the trunk and affected limbs using gentle, rhythmic massage action.
  Interventions: Device: Flexitouch System with Standard Wound Care

INTERVENTIONS:
Device: Standard Wound Care
  Other Names: Farrow Wrap, Acticoat, Aquacel Ag, or Mepilex Ag foam dressings
  Arms: Standard Wound Care
Device: Flexitouch System with Standard Wound Care
  Other Names: Flexitouch system, Farrow Wrap, Acticoat, Aquacel Ag, or Mepilex Ag foam dressings
  Arms: Flexitouch system with Standard Wound Care

SUMMARY:
This is a study to compare the healing process of venous stasis ulcers when the Flexitouch® system is added to the standard treatment of venous ulcers. We hypothesize that adding the Flexitouch® system to standard venous ulcer treatment will result in

1. greater complete healing
2. greater percentage reduction in ulcer area
3. reduced time to complete healing, as compared to the use of standard treatment alone
4. a greater reduction in affected leg volume as compared to standard treatment alone.

DETAILED DESCRIPTION:
A pilot randomized trial of Flexitouch® as an adjunctive treatment for venous ulcers

Objectives To determine if the Flexitouch® compression therapy system, when added to standard venous ulcer (VU) treatment, results in: 1. Greater complete healing at 12 weeks as compared to standard treatment alone. 2. Greater percentage reduction in ulcer area at 12 weeks as compared to standard treatment alone. 3. Less time to complete healing as compared to standard treatment alone 4. A greater reduction in the leg volume of the affected leg

Hypothesis We hypothesize that adding the Flexitouch® system to standard venous ulcer treatment will result in

1) greater complete healing, 2) greater percentage reduction in ulcer area 3) reduced time to complete healing, as compared to the use of standard treatment alone, and 4) a greater reduction in affected leg volume as compared to standard treatment alone.

Patient recruitment, eligibility, and exclusions Patients who present at our clinic with a venous leg ulcer, as judged by clinical presentation and history, will be recruited for participation in this research study. For this pilot study a total of 16 patients will be recruited.

Protocol and Procedures After verifying eligibility and administering an approved informed consent, patients will be randomized to one of the study arms (A or B). Study patients will be seen one or two times per week (per physician's discretion) for 12-weeks for standard wound care and treatment. For both groups, sustained compression will be achieved with the FarrowWrap™ Classic device. This device will be worn continuously except during the twice-weekly treatments and when Flexitouch therapy is being undertaken (Group B only). Group B will use Flexitouch at home every day (twice daily); Group A will not use Flexitouch. Once per week, treatment and parameter assessments will be undertaken as described below.

Standard Wound Care and Treatment Standard wound care treatment will include gentle wound ulcer cleansing with saline solution at each visit, maintaining moisture balance in the wound and periwound with appropriate dressings (e.g Acticoat, Aquacel Ag, or Mepilex Ag foam dressings), reminding subjects of the importance of proper nutrition, leg elevation at rest and activity, including frequent ambulation and ankle range of motion exercises through the day. The FarrowWrap Classic device is applied over the dressing to achieve suitable compression pressures as an important component of the standard treatment. For venous ulcer treatment it is applied at full stretch. The patient will be given instructions as to how to apply the FarrowWrap at home.

Flexitouch System and its Use Patients who have been randomized to Group B will be provided a home Flexitouch unit. They will be given instructions to use it on a twice daily basis. They will be instructed to remove the FarrowWrap during the time they are using Flexitouch. The Flexitouch System works by applying dynamic low-pressure compression to the trunk and affected limbs using gentle, rhythmic massage action. The system consists of a controller unit with four eight-port connectors and a garment set for the trunk and leg. The garments are placed around the trunk and affected limbs and are connected to the controller by a tubing harness. The controller inflates and deflates the air chambers within the garments in a pre-determined pattern to assist the lymphatics in moving the fluid into adjacent lymph node regions of the trunk. The controller inflates individual chambers in the garments for 1-3 seconds per inflation.

Potential Treatment modifications The patient's welfare, as determined by the principal investigator, will take precedence over any study procedures. Any interventions necessary for the patient's welfare will be undertaken as necessary.

Wound Photography The wound will be photographed using a digital camera with zoom capability supplied by the sponsor of this study. All photographs will be taken with the camera pointing directly down to the wound such that the angle between the camera and the plane-of-the wound is as near to 90o as possible. Flash will be avoided if there is adequate lighting. The vertical distance from the wound to the camera is not critical but a distance of about 20 cm will be used when possible. Prior to taking photographs, a suitable dimensional scale or calibration standard will be placed in contact with the skin near, but outside a wound margin. In the case of a one-dimensional scale, it will be placed above or below the wound, and positioned along the long dimension of the wound. A suitable calibration standard will be supplied by the sponsor of this study. The framing of the photo will be such as to include 1) the complete wound bed, 2) a small sampling of the surrounding periwound tissue and 3) the calibration standard or scale. The composed image, as viewed through the camera LCD viewport, will be as large as possible while still including the required elements. The camera will be oriented such that the horizontal dimension of the LCD viewport is parallel to the horizontal calibration scale on the leg.

Wound Tracing After photographing, the wound margins will be traced by placing a transparent grid over the wound. The grid is a commercial product (E-Z Graph) that is designed for this purpose. It consists of two layers; a bottom layer which is in contact with the wound and an upper layer on which tracing is done using a colored pen. The upper layer has a grid system with 1 x 1 cm squares imbedded into the material. After tracing the bottom layer is discarded. The patient's study ID, visit number and visit date are then recorded on a space provided on the upper tracing grid.

Assessment of Leg Volumes Leg volumes of both right and left legs from ankle to knee will be determined. This is done using a calibrated tape measure (Gulick-type) to measure circumferences at 4 cm intervals starting at the malleoulus and progressing toward the knee. From these circumference measurements, limb volumes will be determined using the well established truncated cone model together with a validated software algorithm. Using this method the wound assessor enters the circumferences into a standardized form and the appropriate volumes are automatically determined.

Assessment of Complete Wound Healing At each visit the wound will be carefully inspected by the Principal Investigator and the presence or absence of complete wound healing noted and recorded. For this study, wound healing will be considered to occur when the wound is fully covered with epithelium and there is no drainage. In addition, at each visit, a study-related case report form will be completed by the Principal Investigator to document various clinical features of the wound and to note any relevant study-related actions or events. This form will be embedded within password protected software so that most wound descriptors will be able to be entered and documented with a simple mouse click.

Analysis of Wound Areas and Related Parameters Wound Areas by Photo Images: The digital images of the wound will be coded by the Principal Investigator by suitably renaming each photographic image file with a unique identifier. He will keep a record of these coded file names and the group, patient, and visit date and number to which they correspond. A copy of each image file will be made and stored on a CD. The CD will be sent to a scientific advisor who works with the study sponsor. The advisor will be responsible for the analyses of the images, including the determination of wound areas via computerized planimetry and for subsequent data and statistical analyses. The analyst will blind as to which actual group the images correspond. At the completion of the data acquisition phase of the study, the analyst will be told which images belong to common groups, but he will still not know which of the common groups belong to which arm of the study. He will thus remain blind during the subsequent statistical analyses.

Wound Areas by Tracings: As a complementary comparison approach, wound areas will also be assessed from the wound tracings. The analyst will be supplied with copies of the coded tracings. The tracings will then be scanned and the wound areas determined by computerized digital planimetry as previously described. Areas determined by this method will serve as a check measurement and will be used as a backup in those cases (if any) in which photographic quality is inadequate.

Leg Volumes: In addition to photographs and tracings, the analyst will be supplied with coded electronic copies of the leg circumference forms. This data will be used to determine if, and to what extent, changes in leg volume or edema occur, and if there are differences in these parameters between groups A and B.

Wound Descriptors: A coded electronic version of the case report form, containing wound descriptor parameters data, will be supplied to the analyst. This information will be used primarily in the final analysis to summarize the clinical progression of the wounds.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must be at least 18 years old
2. The ulcer maximum length x its maximum width must be greater or equal to 0 cm2
3. The ulcer must extend through both the epidermis and dermis, with no exposed tendon or bone.
4. The ulcer must have been present for more than 1 month.
5. The ulcer must be located below the knee.
6. The ulcer bed must have some viable tissues with some granulation tissue.

Exclusion Criteria:

1. Exposed bone, tendon, or fascia
2. Severe rheumatoid arthritis
3. History of radiotherapy to the ulcer site
4. Uncontrolled congestive heart failure
5. Receiving corticosteroids or immune suppressive therapy
6. History of collagen vascular disease
7. Known malnutrition (albumin<3.0 g/dL). If malnutrition is suspected, the albumin level should be checked to determine if the patient meets the albumin criterion.
8. The ulcer is clinically infected. However, patients may be entered into the study after successful treatment of infection.
9. Known uncontrolled diabetes (HgbA1c > 8%). If uncontrolled diabetes is suspected, the Hgb A1c should be checked to determine patient eligibility.
10. Signs of cellulitis, osteomyelitis, or necrotic or avascular ulcer bed(s).
11. Known arterial insufficiency (Ankle-brachial index < 0.7, or TcPO2 < 35 mm Hg, or Toe-brachial index < 0.4). If peripheral vascular disease is suspected, vascular lab testing should be checked to determine patient eligibility.
12. Active sickle cell disease
13. Unable to comply with the procedures described in the protocol
14. Enrolled in a clinical evaluation for another investigational wound-care device or drug
15. Patients diagnosed with deep venous thrombosis or phlebitis in the affected limb in the last 6 months
16. Pregnancy, suspected or confirmed
17. Chronic renal disease, if deemed by the principal investigator to be severe enough to interfere with wound healing
18. Known active or recurrent cancer, or currently receiving chemotherapy or radiation therapy
19. History or pulmonary embolism
20. Poorly controlled asthma
21. Pulmonary Edema

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2007-09; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wade Farrow, MD, Principal Investigator — Wound Healing and Hyperbaric Center; Sunday Hoy, JD, Study Director — Tactile Systems Techonology Inc.
Locations (2):
- United States (2):
  - VA Medical Center, Minneapolis, Minnesota
  - Wound Healing and Hyperbaric Center, College Station, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was stopped early due to slow accrual.
Groups:
- Standard of Care: Standard Wound Care using compression
- Flexitouch System: Flexitouch system with Standard Wound Care using compression
Period: Overall Study
Arm/Group | Standard of Care | Flexitouch System
Started | 4 | 4
Completed | 4 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Standard of Care Wound Treatment: Standard Wound Care using compression
- Flexitouch System With Standard of Care: Flexitouch system with Standard Wound Care using compression
- Total: Total of all reporting groups
Arm/Group | Standard of Care Wound Treatment | Flexitouch System With Standard of Care | Total
Number analyzed (Participants) | 4 | 4 | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 3 | 6
  >=65 years | 1 | 1 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 59 (9.8) | 54 (18.9) | 56.5 (14.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 3 | 3 | 6
Region of Enrollment [Number; unit: participants]
  United States | 4 | 4 | 8

OUTCOME MEASURES:

1. Primary Outcome: Wound Healing
Time Frame: 12 weeks
Population: The study was stopped early due to lack of enrollment statistical analysis was not completed.
Arm/Group | Standard of Care Wound Treatment | Flexitouch System With Standard of Care
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Reduction in Leg Volume
Time Frame: 12 weeks
Population: The study was stopped early due to lack of enrollment statistical analysis was not completed.
Arm/Group | Standard of Care Wound Treatment | Flexitouch System With Standard of Care
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Standard of Care Wound Treatment | Flexitouch System With Standard of Care
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4
Other Adverse Events (participants affected / at risk) | 0/4 | 2/4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard of Care Wound Treatment (N=4) | Flexitouch System With Standard of Care (N=4)
Mild urticaria - Allergic reaction to new food (Immune system disorders) | 0 (0) | 1 (1) — Subject experienced mild urticaria after eating. Resolved with medicaiton.
Bruise - red mark on foot from brace (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — The patient expereinced a red mark on their mid foot from the brace they wore on their leg. Investigator felt that this could be possibly related to compression garment,provided additional padding on leg, the event resolved.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less